CLINICAL TRIAL: NCT05892016
Title: Soft Tissue Contour and Radiographic Evaluation of Ridge Preservation Using Different Techniques
Brief Title: Ridge Preservation Using Different Techniques
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Cheng-En Sung, Assistant professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A202305015
Record Dates: First submitted 2023-05-02; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Alveolar Ridge Augmentation; Connective Tissue; Tooth Extraction; Membranes; Retained
Keywords: Alveolar Ridge Preservation Connective tissue graft; Tooth extraction; Membranes

STUDY DESIGN:
Intervention Model Description: 1. spontaneous healing (control) Alveolar ridge preservation grafted with bone particle and
  2. covered with a free palatal graft
  3. covered with pedical palatal graft
  4. covered with a collagen membrane
  5. covered with a non-resorbable high-density polytetrafluoroethylene membrane.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- spontaneous healing (No Intervention): No treatment after tooth extraction
- Bone particle + subepithelial connective tissue graft (Experimental): Alveolar ridge preservation grafted with bone particle and covered with a subepithelial connective tissue graft
  Interventions: Procedure: Alveolar ridge preservation
- Bone particle + Vascularized interpositional periosteal connective tissue graft (Experimental): Alveolar ridge preservation grafted with bone particle and covered with vascularized interpositional periosteal connective tissue graft
  Interventions: Procedure: Alveolar ridge preservation
- Bone particle + collagen membrane (Experimental): Alveolar ridge preservation grafted with bone particle and covered with a collagen membrane
  Interventions: Procedure: Alveolar ridge preservation
- Bone particle + Cytoplast (Experimental): Alveolar ridge preservation grafted with bone particle and covered with a Cytoplast.
  Interventions: Procedure: Alveolar ridge preservation

INTERVENTIONS:
Procedure: Alveolar ridge preservation — grafted with bone particle and covered with a subepithelial connective tissue graft
  Arms: Bone particle + Cytoplast; Bone particle + Vascularized interpositional periosteal connective tissue graft; Bone particle + collagen membrane; Bone particle + subepithelial connective tissue graft
Procedure: Alveolar ridge preservation — grafted with bone particle and covered with vascularized interpositional periosteal connective tissue graft
  Arms: Bone particle + Cytoplast; Bone particle + Vascularized interpositional periosteal connective tissue graft; Bone particle + collagen membrane; Bone particle + subepithelial connective tissue graft
Procedure: Alveolar ridge preservation — grafted with bone particle and covered with a collagen membrane
  Arms: Bone particle + Cytoplast; Bone particle + Vascularized interpositional periosteal connective tissue graft; Bone particle + collagen membrane; Bone particle + subepithelial connective tissue graft
Procedure: Alveolar ridge preservation — grafted with bone particle and covered with a Cytoplast
  Arms: Bone particle + Cytoplast; Bone particle + Vascularized interpositional periosteal connective tissue graft; Bone particle + collagen membrane; Bone particle + subepithelial connective tissue graft

SUMMARY:
Soft tissue contour and radiographic evaluation of alveolar ridge preservation using different techniques

Background:

Following tooth extraction, the alveolar ridge undergoes an inevitable remodeling process which influences future implant therapy or prosthetic rehabilitation in the edentulous area. In an attempt to attenuate the loss of hard and soft tissue after tooth loss, alveolar ridge preservation (ARP) immediately after complete tooth extraction could minimize the need for ancillary ridge augmentation or soft tissue grafting. Different techniques and barrier membranes has been proposed to achieve the sealing of extraction socket.

Aim:

To investigate the effect of different techniques and barrier membranes for the soft tissue contour and morphological change of alveolar ridge after ARP

Methods:

The study was designed as a randomized controlled trial and recruited patients, who require ARP for the purpose of implant placement or prosthodontic rehabilitation. After the tooth extraction, patients were randomly allocated to one of the following groups: ridge preservation with a xenogeneic bone substitute and (a) spontaneous healing (control), (b) covered with a free palatal graft, (c) or covered with pedical palatal graft, (d) covered with a collagen membrane, (e) covered with a non-resorbable high-density polytetrafluoroethylene membrane. 2 weeks, 4 weeks, 12 weeks, and 24 weeks following tooth extraction and ARP, clinical profilometric and radiographic evaluations were performed to analyze the change of hard and soft tissue contour. Moreover, and the need for additional guided bone regeneration (GBR) or soft tissue augmentation were assessed prior implants or fixed prosthesis placement.

ELIGIBILITY:
Inclusion Criteria:

* >20 years old
* No contraindications for invasive dental procedures.
* Not pregnant.
* Teeth need to be extracted due to malocclusion or broken teeth.
* Requires dental implant or denture fabrication after tooth extraction.
* Healthy soft tissue (probing bleeding index <20%, plaque index <20%).
* At least 2mm of keratinized gingiva on the buccal and lingual sides.
* No need for simultaneous bone augmentation surgery during implant placement.
* Willing to participate in and sign the consent form for this trial.

Exclusion Criteria:

* Poor oral hygiene maintenance.
* Uncontrolled periodontal disease.
* Heavy smoker (smokes >20 cigarettes per day).
* Uncontrolled diabetes.
* Alcohol abuse.
* Currently receiving medication treatment affecting wound healing (osteoporosis medication, radiation or chemotherapy).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Soft tissue alternation | up to 12 months
  cone-beam computed tomography data and STereoLithography files are superimposed to measure the soft tissue dimensions.
Hard tissue alternation | up to 12 months
  cone-beam computed tomography data and STereoLithography files are superimposed to measure the hard tissue dimensions.

SECONDARY OUTCOMES:
Keratinized tissue width changes | up to 12 months
  Use periodontal probe to measurement.
Visual Analogue Scale | 14 days
  Ask the patient to fill out the questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No